CLINICAL TRIAL: NCT01946698
Title: A Study on the Differences in Inflammatory Markers Between Women With Endometriosis and Women Without in Relation to Fertility and Food Consumption.
Brief Title: Endometriosis, Food Consumption and Fertility
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Ulla Breth Knudsen, Professor, Consultant, Ph.D., University of Aarhus
Other Study IDs: Endo
Record Dates: First submitted 2013-08-18; First posted 2013-09-20 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Biospecimen Retention: Samples With DNA — Blood samples for inflammatory markers, hormones and genetic testing. Follicular fluid for inflammatory markers. Cells from the uterus for testing of different additives and what characterize cells from women with endometriosis compared to controls.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fertility patients: Women with endometriosis compared to women without endometriosis. Different samples will be collected (blood, follicular fluid, cells from the uterus)

SUMMARY:
To investigate parameters related to fertility in women with endometriosis in relation to food items.

DETAILED DESCRIPTION:
The study has been reviewed and accepted by the legal registrations in Denmark (The Regional Committee on Biomedical Research Ethics and The Danish Dataprotection Agency). The data will be anonymous and kept as described by the Danish register law.

ELIGIBILITY:
Inclusion Criteria:

* Fertility patients

Exclusion Criteria:

* mental challenges

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women attending an infertility Clinic, some with endometriosis compared to women without endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-12 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
The level of Free Fatty Acid in follicular fluid will be different in women with endometriosis compared to controls | The fluid will be collected, frozen and tested december 2014

SECONDARY OUTCOMES:
methylation pattern of specific genes in the endometrium | Collecting of cells and testing december 2014
  The cells will be collected from infertile women with or without endometriosis, frozen and tested later.

CONTACTS AND LOCATIONS:
Overall Officials: Ulla B Knudsen, Professor, Principal Investigator — Professor, Consultant at the Fertility Clinic, Arhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark